CLINICAL TRIAL: NCT00762697
Title: Obtaining and Storing Blood Samples and Debridement Samples for Wound Related Research
Status: Completed | Type: Observational
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Principal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-006
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Venous Insufficiency
Keywords: diabetic, venous insufficiency
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Analytical methods used to examine the blood or debridement can investigate morphological, molecular, immunological, cellular, viral, biochemical, chemical, genetic, and/or transcriptional components of the samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The intent of this protocol is to obtain blood samples from subjects with or without a wound, so the blood can be used in wound-related scientific studies. It is also the intent of this protocol to salvage debrided wound material that is normally destined for destruction, so it can be used in wound-related scientific studies.

DETAILED DESCRIPTION:
The samples will be studied in order to attempt to better understand wounds and their associated barriers to healing. Analytical methods used to examine the blood or debridement can investigate morphological, molecular, immunological, cellular, viral, biochemical, chemical, genetic, and/or transcriptional components of the samples. It is the goal of this study to determine if these tests may be able to provide important insights into the keys of wound healing, wound persistence, or wound deterioration.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for the Collection of Wound Debridement

1. The subject must have a full thickness wound.
2. The subject must be a candidate for sharp debridement.
3. The subject must be 18 years of age or older.
4. The subject must be mentally competent as determined by the Investigator Inclusion Criteria for the Collection of Blood

Wounded or Otherwise Not Healthy Subjects, Subjects Weighing Less Than 110 lbs., or Subjects Contributing 50ml of Blood or Less:

1. The subject must be 18 years of age or older.
2. The subject must be mentally competent as determined by the Investigator.

Not Wounded and Healthy Subjects Weighing at Least 110 lbs. Who May Contribute Up To 500ml of Blood:

1. The subject must be 18 years of age or older.
2. The subject must be mentally competent as determined by the Investigator.
3. The subject must weigh at least 110 lbs.
4. The subject must have a hemoglobin level that is in or above the normal range within the last 8 (eight) weeks as determined by standard clinical laboratory testing, the copper sulfate test, or a point of care instrument.

Exclusion Criteria:

Exclusion Criteria for the Collection of Wound Debridement and Blood Collection*

1. The subject must not be currently incarcerated or pregnant.
2. The subject must not weigh less than 40 lbs.
3. If the subject will be contributing more that 50 ml of blood during an 8 (eight) week period, then the subject must not have donated red blood cells within the last 8 (eight) weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with venous insufficiency, diabetic foot ulcers, decubitus ulcers.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Wolcott, MD, Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States